CLINICAL TRIAL: NCT01351038
Title: A Two Stage Multicenter Phase II Trial of Concurrent Induction Chemoimmunotherapy With Epirubicine, Oxaliplatin, Capecitabine and Panitumumab in KRAs Wild-type, Resectable Type II Gastric Adenocarcinoma
Brief Title: Concurrent Induction Chemoimmunotherapy With Epirubicine, Oxaliplatin, Capecitabine and Panitumumab in KRAs Wild-type, Resectable Type II Gastric Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: REAL trial showed a significant difference in OS for reduced EOX and standard EOX
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Amgen (Industry)
Responsible Party: Dr. Daniela Wolkersdorfer, Arbeitsgemeinschaft für medikamentöse Tumortherapie GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT Gastric-4
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: KRAS Wild Type; Resectable Type II Gastric Adenocarcinoma
MeSH Terms: interventions — Epirubicin; Oxaliplatin; Capecitabine; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): 3 cycles(repeated q21d) Epirubicine 50mg/m² i.v. d1 Oxaliplatin 100mg/m² i.v. d1 Capecitabine 500mg/m² bid d1-d21 Panitumumab 9mg/kg i.v. d1
  Interventions: Drug: Epirubicine, Oxaliplatin, Capecitabine, Panitumumab

INTERVENTIONS:
Drug: Epirubicine, Oxaliplatin, Capecitabine, Panitumumab — 3 cycles (repeated q 21d) Epirubicine 50mg/m² i.v. d1 Oxaliplatin 100mg/m² i.v. d1 Panitumumab 9mg/kg i.v. d1 Capecitabine 500mg/m² bid d1-21

SUMMARY:
This is an open label, multicenter, single-arm phase II trial with primary eqirubicine-oxaliplatin-capecitabine chemotherapy and concurrent Pmab in patients with resectable, histologically proven gastric or esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Untreated, histologically confirmed, KRAS wild type, resectable gastric or esophageal adenocarcinoma
* T2-4 NX M0 disease
* ECOG performance status 0-1
* adequate hematological status
* adequate renal function
* adequate hepatic function
* adequate metabolic function

Exclusion Criteria:

* pregnant or breast feeding women
* previous malignancy other than gastric cancer in the last 5 years except curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix
* arterial or venous thromboembolism within 6 months before enrollment
* clinically significant cardiovascular disease within 1 year before enrollment
* history of interstitial lung disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)

PRIMARY OUTCOMES:
Efficacy
  Proportion of patients with T0 ant T1 disease after neoadjuvant combined chemoimmunotherapy
Safety
  Proportion of patients with grade 4 diarrhea

SECONDARY OUTCOMES:
Histopathological response
  rate of complete pathological response
overall survival after one year
Progression free survival after one year
Proportion of patients completing 3 treatment cycles
Safety
  NCI CTCAE v.3

CONTACTS AND LOCATIONS:
Locations (6):
- Austria (6):
  - LKH Feldkirch, Feldkirch
  - KH Elisabethinen Linz, Linz
  - AKh Linz, Linz
  - Universitätsklinik für Innere Medizin III, Salzburg
  - Klinikum Kreuzschwestern Wels GmbH, Wels
  - St. Vinzenz Krankenhaus Betriebs GmbH, Zams